CLINICAL TRIAL: NCT05640219
Title: Benha Modification for Renal Track Creation in Percutaneous Nephrolithotomy (PCNL), How and Why?
Brief Title: Novel Technique for PCNL Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Collaborators: mohamed abdelzaher (Unknown)
Responsible Party: Principal Investigator, mohamed abdelrahman alhefnawy, assistant professor, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PCNL track
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: PCNL
Keywords: complications, partial staghorn stones, PCNL

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: laparoscopic trocar 12mm — long laparoscopic trocar 12mm (36 french) with central hole from its tip till its handle with transparent sheath

SUMMARY:
Benha modification for renal track creation in percutaneous nephrolithotomy (PCNL) Our modification aims to decrease the complications of PCNL in large stones

DETAILED DESCRIPTION:
Introduction : PCNL occupies the best stone management modality till now in large stones with promissing impacts as regard to morbidity and hospital stay time. (1,2,3) Many reported complications due to PCNL either intra or postoperative especially in large stones up to 83% including bleedng and extravasation .(4) Single step dilatation during PCNL track forminghave many advantages over sequential dilatation as it ismore economic with less blood loss and less radiation exposure, so it is advantageous than conventional Alken or teflon sequential dilators also it is more economic than balloon dilators. (5,6,7,8) To decrease the incidence bleeding, the manipulation should be limited and transpapillary puncture should be kept. (9) Extravasation remains one of the most serious complication during PCNL as vigorousabsorption of the irrigant fluid may cause electrolyte disbalance that may lead to cardiac complications (overload) or brain edema.. (10) Objective : Our modification aims to decrease the complications of PCNL in large stones.

Patients and methods : Our modification will be performed in our department in Benha univerisity hospital with a written consent on 10 patients with partial staghorn stone more than 4 cm occupying the renal pelvis and the lower calyx +/_ the upper calyx in patints 18 years old or more. Also, patients with uncorrected bleeding disorders, moderate or high risk cardiac patients , active urinary tract infection , skletal deformities or patients with complete staghorn stone will be excluded.

Preoperative assesment:

* full history and clinical examination
* full laboratory investigation including heamoglobin (Hb) and serum creatinine (Scr)
* radiological investigation as pelviabdomenal ultrasound , plain X ray (KUB) and coputerized tomography (CT)

Intraoperative assesment:

Under general anaesthesia, after ureteric catheter insertion and using fluoroscopic guidancein prone position introducing a superstiff guide wire targeting the posterior lower calyx transpapillary by puncture needle application then by a straight long artery beside the puncture needle advancing it till penetrating the fascia then open it in two different perpendicular planes to creat a wide tract permitting single step dilatation over the stiff guide wire then safety guide wire will be inserted .Using a long laparoscopic trocar 12mm (36 french) with central hole from its tip till its handle with transparent sheath also a side scrow included to adjust the irrigation fluid outflow and permitting using a suction system if stone disintegration performed while saline irrigation through the ureteric catheter was acting.

The superstiff wire will pass through the tip hole of the trocar ,then under C arm imaging the trocar directed to the targeted calx transpapillary not reaching the calyceal neck then nephroscopy and pneumatic lithotripsy used and then large fragments will be extracted and may reaches 1.5 to 2 cm.

Till the procedure end ,intraoperative time and the need for blood transfusion will be recorded.

Nephrotomy tube 28 f will be fixed in all cases.

Postoperative assessment:

Postoperative Hb , Scr KUB and CT if needed in the next morning will be performed, Also hospital stay and postoperative complications will be registered as fever , heamaturia and leakage from the nephrostoy tube site after its removal.

Keywords: single step dilatation, complications, partial staghorn stones, percutaneous nephrolithotomy Financial support and sponsorship Nil. Conflicts of interest There are no conflicts of interest.

References :

1. Geraghty J.P. and Somani B.K. (2017): Worldwide Trends of urinary stone disease treatment over the last two decades: a systematic review. J Endourol.; 31(6):547-556.
2. Jones P., Elmussareh M., Aboumarzouk O. M., Mucksavage P. and Somani B. K.(2018): Role of Minimally Invasive (Micro and Ultra-mini) PCNL for Adult Urinary Stone Disease in the Modern Era: Evidence from a Systematic Review. Current Urology Reports 19: 27.
3. Turk C, Petrik A, Sarica K, Seitz C, Skolarikos A, Straub M,Drake T ,Donaldson JF ,and Rubayel L (2019): EAU guideline on urolithiasis. [Accessed 2 July 2019]
4. Michel MS, Trojan L,and Rassweiler JJ(2007): Complications in Percutaneous Nephrolithotomy in European urology.; 51(4)899-906.
5. El-Shazly M, Salem S, Allam A, Hathout B. Balloon dilator versus telescopic metal dilators for tract dilatation during percutaneous nephrolithotomy for staghorn stones and calyceal stones. Arab J Urol 2015;13:80-3.
6. Nour HH, Kamal AM, Zayed AS, Refaat H, Badawy MH, El-Leithy TR, et al. Single-step renal dilatation in percutaneous nephrolithotomy: A prospective randomised study. Arab J Urol 2014;12:219-22.
7. Suelozgen T, Isoglu CS, Turk H, Yoldas M, Karabicak M, Ergani B, et al. Can we use single-step dilation as a safe alternative dilation method in percutaneous nephrolithotomy? Urology 2017;99:38-41.
8. Desai MR, Sharma R, Mishra S, Sabnis RB, Stief C, Bader M, et al. Single-step percutaneous nephrolithotomy (microperc): The initial clinical report. J Urol 2011;186:140-5.
9. Akman T, Binbay M, Sari E, Yuruk E, Tepeler A, Akcay M,Muslumanoglu AY and Tefekli.A (2011). Factors affecting bleeding during percutaneousnephrolithotomy: single surgeon experience. J Endourol; 25:327e33
10. Taylor E, Miller J, Chi T,and Stoller ML (2012). Complications associated with percutaneous nephrolithotomy. Transl Androl Urol ; 1:223-228.

ELIGIBILITY:
Inclusion Criteria:

patients with partial staghorn stone more than 4 cm occupying the renal pelvis and the lower calyx +/_ the upper calyx in patints 18 years old or more

Exclusion Criteria:

patients with uncorrected bleeding disorders, moderate or high risk cardiac patients , active urinary tract infection , skletal deformities or patients with complete staghorn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2023-03-07 (Estimated); Study Completion 2023-03-17 (Estimated)

PRIMARY OUTCOMES:
decrease the intraoperative complication | intraoperative
  assessing the operative time in minutes
blood loss in the operative theatre | intraoperative
  pre and postoperative haemoglobine in gram/dl

SECONDARY OUTCOMES:
early postoperative impact and incidence of complication | withen 10 days postoperative
  fever, heamaturia and leakage from the nephrostomy site